CLINICAL TRIAL: NCT00378079
Title: Methadone Maintenance for Prisoners
Acronym: MMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA016237-03 (NIH); R01DA016237 (NIH)
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Heroin Addiction
MeSH Terms: conditions — Heroin Dependence | interventions — Counseling; Parturition; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 (Experimental)
  Interventions: Drug: Counseling + Methadone
- 1 (Active Comparator)
  Interventions: Other: Counseling Only
- 2 (Experimental)
  Interventions: Drug: Counseling + Transfer

INTERVENTIONS:
Other: Counseling Only — Counseling only in prison, with passive referral to drug abuse treatment upon release
  Arms: 1
Drug: Counseling + Transfer — Counseling only in prison, with opportunity to enter methadone maintenance upon release
  Arms: 2
Drug: Counseling + Methadone — Counseling and methadone maintenance in prison, with opportunity to continue that treatment upon release
  Arms: 3

SUMMARY:
This five-year study examines the benefits of methadone maintenance treatment initiated in prison and continued in the community to male offenders who were previously, but not currently, heroin-dependent. It is anticipated that such prisoners will have more favorable outcomes in the year following release with regard to drug abuse, crime, and HIV risk behavior than either prisoners who receive counseling only or begin initiation of methadone maintenance in the community

DETAILED DESCRIPTION:
Most prisoners with histories of pre-incarceration heroin addiction do not receive treatment while incarcerated or upon release. Effective treatment for such prisoners is urgently needed because rapid relapse typically follows release. Relapse is associated with increased risk for HIV, overdose death, criminal activity, and reincarceration. Other than three studies of methadone maintenance with short-term jail inmates, the only study of longer-term inmates who were previously, but not currently, heroin-dependent was the investigator's pilot study with pre-release inmates. Based on that pilot study, which found that initiating maintenance treatment is feasible and facilitates post-release treatment entry, the present study provides a more rigorous examination of this unique treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Heroin dependence in the year prior to current incarceration
* 3-6 months left to serve in prison-male pre-release inmate suitability for methadone maintenance as determined by medical evaluation
* Willingness to enroll in methadone maintenance
* Having a Baltimore address

Exclusion Criteria:

* Pending parole hearing
* Pending charges
* Kidney failure
* Liver failure

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2003-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Kinlock, Ph.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Metropolitan Transition Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kinlock TW, Schwartz RP, Gordon MS. The significance of interagency collaboration in developing opioid agonist programs for inmates. Corrections Compendium 30(3)6-9,28-30,2005.
- [Result] Kinlock TW, Gordon MS, Schwartz RP, O'Grady K, Fitzgerald TT, Wilson M. A randomized clinical trial of methadone maintenance for prisoners: results at 1-month post-release. Drug Alcohol Depend. 2007 Dec 1;91(2-3):220-7. doi: 10.1016/j.drugalcdep.2007.05.022. Epub 2007 Jul 12. PMID 17628351
- [Result] Kinlock TW, Gordon MS, Schwartz RP, O'Grady KE. A Study of Methadone Maintenance For Male Prisoners: 3-Month Postrelease Outcomes. Crim Justice Behav. 2008;35(1):34-47. doi: 10.1177/0093854807309111. PMID 18612373
- [Result] Gordon MS, Kinlock TW, Schwartz RP, O'Grady KE. A randomized clinical trial of methadone maintenance for prisoners: findings at 6 months post-release. Addiction. 2008 Aug;103(8):1333-42. doi: 10.1111/j.1360-0443.2008.002238.x. PMID 18855822
- [Result] Kinlock TW, Gordon MS, Schwartz RP, Fitzgerald TT, O'Grady KE. A randomized clinical trial of methadone maintenance for prisoners: results at 12 months postrelease. J Subst Abuse Treat. 2009 Oct;37(3):277-85. doi: 10.1016/j.jsat.2009.03.002. Epub 2009 Mar 31. PMID 19339140
- [Result] Wilson ME, Kinlock TW, Gordon MS, O'Grady KE, Schwartz RP. Postprison release HIV-risk behaviors in a randomized trial of methadone treatment for prisoners. Am J Addict. 2012 Sep-Oct;21(5):476-87. doi: 10.1111/j.1521-0391.2012.00250.x. PMID 22882399
- [Result] Kinlock TW, Gordon MS, Schwartz RP, O'Grady KE. Individual Patient and Program Factors Related to Prison and Community Treatment Completion in Prison-Initiated Methadone Maintenance Treatment. J Offender Rehabil. 2013 Oct;52(8):509-528. doi: 10.1080/10509674.2013.782936. PMID 25580067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: See publication in Journal of Substance Abuse Treatment (2009), 37, 277-285.In summary, participants were recruited between September 2003 and June 2005 from male prisoners in a Baltimore pre-release facility. They had to have met criteria for methadone maintenance treatment in the year prior to incarceration.
Pre-assignment Details: See above
Groups:
- 1 Counseling Only in Prison: Counseling Only : Counseling only in prison, with passive referral to drug abuse treatment upon release
- 2 Counseling Only in Prison, With Initiation of Methadone Main: Counseling + Transfer : Counseling only in prison, with opportunity to enter methadone maintenance upon release
- 3 Counseling and Methadone Maintenance in Prison, With Continu: Counseling + Methadone : Counseling and methadone maintenance in prison, with opportunity to continue that treatment upon release
Period: Overall Study
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Started | 70 | 70 | 71
Completed | 64 | 69 | 71
Not Completed | 6 | 1 | 0
Not completed — Lost to Follow-up | 6 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu | Total
Number analyzed (Participants) | 70 | 70 | 71 | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 71 | 211
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (7.5) | 40.3 (6.7) | 39.9 (7.0) | 40.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 70 | 70 | 71 | 211
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 71 | 211

OUTCOME MEASURES:

1. Primary Outcome: Treatment Retention in the Community
Description: days in community treatment
Time Frame: one year post prison release
Measure: Mean (Standard Deviation); unit: Days in community treatment
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Number analyzed (Participants) | 64 | 69 | 71
Days in community treatment | 23.1 (72.5) | 91.3 (144.6) | 166.0 (166.4)

2. Primary Outcome: Heroin Use
Description: opioid urine test results-percent of participants who were opioid-positive
Time Frame: results at one year post prison release
Population: Includes participants who provided urine samples at the time their 1-year post-prison release assessment was due-excludes those assessed later or reincarcerated
Measure: Number; unit: % participants opioid positive
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Number analyzed (Participants) | 32 | 39 | 44
% participants opioid positive | 65.6 | 48.7 | 25.0

3. Primary Outcome: Cocaine Use
Description: cocaine urine test results-percent of participants testing positive for cocaine
Time Frame: one year post prison release
Population: Includes participants who provided urine samples at the time their 1-year post-prison release assessment was due, excludes those assessed later or reincarcerated
Measure: Number; unit: percent cocaine positive participants
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Number analyzed (Participants) | 32 | 39 | 44
percent cocaine positive participants | 71.9 | 66.6 | 43.2

4. Primary Outcome: HIV-risk Behaviors
Time Frame: one year
Reporting Status: Not Posted

5. Primary Outcome: Criminal Activity
Description: self reported days of criminal activity
Time Frame: one year post prison release
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Number analyzed (Participants) | 64 | 69 | 71
number of days | 106.7 (128.7) | 65.2 (96.2) | 81.8 (109.5)

6. Secondary Outcome: Employment
Description: number of days employed, past 30 days-self report, assessed one year post-prison release
Time Frame: one year
Measure: Mean (Standard Deviation); unit: number of days employed, past 30
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Number analyzed (Participants) | 64 | 69 | 71
number of days employed, past 30 | 12.0 (10.3) | 10.3 (10.9) | 8.5 (10.5)

ADVERSE EVENTS:
Time Frame: at any time up to one year after release from prison
Description: The first series of results reports the number and percent of participants by treatment condition who died. The second series involve hospitalizations-the number of participants in each condition that had one or more hospitalizations and the number of events. Other (non-serious) Adverse Events were not collected/assessed..
Arm/Group | 1 Counseling Only in Prison | 2 Counseling Only in Prison, With Initiation of Methadone Main | 3 Counseling and Methadone Maintenance in Prison, With Continu
Serious Adverse Events (participants affected / at risk) | 15/70 | 6/70 | 16/71
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Counseling Only in Prison (N=70) | 2 Counseling Only in Prison, With Initiation of Methadone Main (N=70) | 3 Counseling and Methadone Maintenance in Prison, With Continu (N=71)
Death (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 1 (1)
hospitalizations (General disorders) | 9 (9) | 5 (14) | 15 (20)

LIMITATIONS AND CAVEATS:
See 2009 manuscript published in the Journal of Substance Abuse Treatment for the a discussion of study limitations. The study was conducted only on males from Baltimore. For results regarding HIV risk behaviors see manuscript by Wilson et. al.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No